CLINICAL TRIAL: NCT07384858
Title: Effects of Attentional Focus Strategies During Isokinetic Quadriceps Training on Strength and Functional Performance in Individuals With Patellofemoral Pain Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seda Ateş, physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/714
Record Dates: First submitted 2025-12-17; First posted 2026-02-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Patellofemoral Pain, PFP
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal focus (Experimental)
  Interventions: Other: Internal focus group
- External focus (Experimental)
  Interventions: Other: External focus

INTERVENTIONS:
Other: Internal focus group — Internal focus refers to directing attention to one's own body movements or muscle activity while performing a task (e.g., focusing on contracting a specific muscle). During isokinetic strength exercises, this group is instructed with commands such as: "Tighten your quadriceps" and "Straighten your knee."
  Arms: Internal focus
Other: External focus — External focus refers to directing attention to the effect of a movement on the environment or an external object, rather than on the body itself. During isokinetic exercise, this group is given the instruction: "Increase and maintain the performance indicator on the screen."
  Arms: External focus

SUMMARY:
Patellofemoral pain syndrome (PFPS) is a multifactorial musculoskeletal condition that is common particularly among young and physically active individuals, negatively affecting activities of daily living and physical performance. Although exercise therapy is considered the gold standard in the management of PFPS, there is limited evidence regarding the effectiveness of motor learning strategies applied during exercise. This study aims to shed light on how motor learning approaches can be optimized in clinical rehabilitation by comparing the effects of internal and external focus strategies used during exercise on muscle activation, functional performance, and pain.

This research will make a methodological contribution to the literature through the objective evaluation of muscle mechanical properties using isokinetic assessment and the MyotonPRO device. The findings are expected to clarify the effects of attentional focus strategies on therapeutic outcomes in PFPS rehabilitation and have the potential to provide an evidence-based guide for physiotherapy practice. In this way, the study may contribute to the development of new approaches aimed at improving both clinical effectiveness and patient adherence.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years.
* Diagnosed with patellofemoral pain syndrome (PFPS).
* Anterior or retropatellar knee pain persisting for at least four weeks with a VAS score > 3.
* Pain exacerbated by at least two functional activities (e.g., squatting, stair climbing, prolonged sitting).
* Willing to regularly participate in the 6-week program throughout the study period.

Exclusion Criteria:

* History of patellar subluxation or dislocation.
* Anterior or posterior cruciate ligament insufficiency.
* Lower extremity fractures.
* Neurological or systemic musculoskeletal disorders.
* Rheumatoid arthritis or other inflammatory joint diseases.
* History of knee surgery, meniscal injury, or any other underlying musculoskeletal condition that would prevent the participant from performing the exercises.
* Pregnancy or postpartum period.
* Participation in a similar exercise program within the last 3 months.
* Radiographic evidence of osteoarthritis classified as Kellgren-Lawrence grade 2 or higher.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Kujala Patellofemoral Pain Score | baseline
  Kujala Patellofemoral Pain Score is a valid and reliable self-reported outcome measure specific to patellofemoral pain syndrome that assesses knee function and pain-related limitations during daily activities.
  The total score ranges from 0 to 100, with higher scores indicating better knee function and fewer symptoms.
Kujala Patellofemoral Pain Score | Week 3 of the Treatment
  Kujala Patellofemoral Pain Score is a valid and reliable self-reported outcome measure specific to patellofemoral pain syndrome that assesses knee function and pain-related limitations during daily activities.
  The total score ranges from 0 to 100, with higher scores indicating better knee function and fewer symptoms.
Kujala Patellofemoral Pain Score | Week 6 of the Treatment
  Kujala Patellofemoral Pain Score is a valid and reliable self-reported outcome measure specific to patellofemoral pain syndrome that assesses knee function and pain-related limitations during daily activities.
  The total score ranges from 0 to 100, with higher scores indicating better knee function and fewer symptoms.

SECONDARY OUTCOMES:
Visual Analog Scale | baseline
  Visual Analog Scale (VAS) is a simple and reliable tool used to assess the intensity of knee pain. Participants rate their pain on a 0 to 10 cm scale, with higher scores indicating greater pain severity. It was used to evaluate changes in pain before and after exercise.
Visual Analog Scale | Week 3 of the Treatment
  Visual Analog Scale (VAS) is a simple and reliable tool used to assess the intensity of knee pain. Participants rate their pain on a 0 to 10 cm scale, with higher scores indicating greater pain severity. It was used to evaluate changes in pain before and after exercise.
Visual Analog Scale | Week 6 of the Treatment
  Visual Analog Scale (VAS) is a simple and reliable tool used to assess the intensity of knee pain. Participants rate their pain on a 0 to 10 cm scale, with higher scores indicating greater pain severity. It was used to evaluate changes in pain before and after exercise.
Isokinetic Muscle Strength Assessment (Isoforce) | baseline
  Muscle performance will be objectively evaluated by measuring concentric strength values of the quadriceps muscle.
Isokinetic Muscle Strength Assessment (Isoforce) | Week 3 of the Treatment
  Muscle performance will be objectively evaluated by measuring concentric strength values of the quadriceps muscle.
Isokinetic Muscle Strength Assessment (Isoforce) | Week 6 of the Treatment
  Muscle performance will be objectively evaluated by measuring concentric strength values of the quadriceps muscle.
Muscle Tone | baseline
  Muscle tone was assessed using the MyotonPRO device, expressed in Hertz (Hz), with higher values indicating increased resting muscle tone.
Muscle Tone | Week 3 of the Treatment
  Muscle tone was assessed using the MyotonPRO device, expressed in Hertz (Hz), with higher values indicating increased resting muscle tone.
Muscle Tone | Week 6 of the Treatment
  Muscle tone was assessed using the MyotonPRO device, expressed in Hertz (Hz), with higher values indicating increased resting muscle tone.
Muscle Stiffness | baseline
  Muscle stiffness was measured using the MyotonPRO device, expressed in Newton per meter (N/m), with higher values indicating greater muscle stiffness.
Muscle Stiffness | Week 3 of the Treatment
  Muscle stiffness was measured using the MyotonPRO device, expressed in Newton per meter (N/m), with higher values indicating greater muscle stiffness.
Muscle Stiffness | Week 6 of the Treatment
  Muscle stiffness was measured using the MyotonPRO device, expressed in Newton per meter (N/m), with higher values indicating greater muscle stiffness.
Muscle Elasticity | baseline
  Muscle elasticity was evaluated using the MyotonPRO device, expressed as logarithmic decrement, with lower values indicating better elastic properties.
Muscle Elasticity | Week 3 of the Treatment
  Muscle elasticity was evaluated using the MyotonPRO device, expressed as logarithmic decrement, with lower values indicating better elastic properties.
Muscle Elasticity | Week 6 of the Treatment
  Muscle elasticity was evaluated using the MyotonPRO device, expressed as logarithmic decrement, with lower values indicating better elastic properties.
Step-Down Test | baseline
  Step-Down Test was used to assess lower-extremity control and functional performance. Participants were instructed to perform as many step-down repetitions as possible within 30 seconds. Performance was recorded as the number of completed repetitions, with higher scores indicating better functional capacity and dynamic knee stability.
Step-Down Test | Week 3 of the Treatment
  Step-Down Test was used to assess lower-extremity control and functional performance. Participants were instructed to perform as many step-down repetitions as possible within 30 seconds. Performance was recorded as the number of completed repetitions, with higher scores indicating better functional capacity and dynamic knee stability.
Step-Down Test | Week 6 of the Treatment
  Step-Down Test was used to assess lower-extremity control and functional performance. Participants were instructed to perform as many step-down repetitions as possible within 30 seconds. Performance was recorded as the number of completed repetitions, with higher scores indicating better functional capacity and dynamic knee stability.
Single-Leg Hop Test | baseline
  Single-Leg Hop Test was used to assess functional performance and dynamic knee stability. Participants were instructed to perform a maximal forward hop on the affected limb. The hop distance was measured in centimeters (cm), with greater distances indicating better functional performance.
Single-Leg Hop Test | Week 3 of the Treatment
  Single-Leg Hop Test was used to assess functional performance and dynamic knee stability. Participants were instructed to perform a maximal forward hop on the affected limb. The hop distance was measured in centimeters (cm), with greater distances indicating better functional performance.
Single-Leg Hop Test | Week 6 of the Treatment
  Single-Leg Hop Test was used to assess functional performance and dynamic knee stability. Participants were instructed to perform a maximal forward hop on the affected limb. The hop distance was measured in centimeters (cm), with greater distances indicating better functional performance.

CONTACTS AND LOCATIONS:
Overall Officials: SEZEN KARABÖRKLÜ ARGUT, Assistant Professor, Study Director — Istanbul University-Cerrahpaşa, Faculty of Health Science
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided